CLINICAL TRIAL: NCT02723578
Title: A Phase 2 Study of Pemetrexed and Erlotinib for Metastatic Colorectal Cancer Refractory to Standard Chemotherapy
Brief Title: Pemetrexed and Erlotinib for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Joong Bae Ahn, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0617
Record Dates: First submitted 2016-03-09; First posted 2016-03-30 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed and Erlotinib (Experimental): Pemetrexed 500 mg/m2 IV over 10 minutes on day 1 every 21 days and Erlotinib 150 mg PO once daily on days 1-21 every 21 days
  Interventions: Drug: Pemetrexed; Drug: Erlotinib

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV over 10 minutes on day 1 every 21 days
Drug: Erlotinib — Erlotinib 150 mg PO once daily on days 1-21 every 21 days

SUMMARY:
Pemetrexed is a multitargeted antifolate, which primarily inhibits thymidylate synthase, dihydrofolate reductase, and glycinamide ribonucleotide formyltransferase in the folate-dependent metabolic process. Nowadays, pemetrexed is used to treat malignant pleural mesothelioma and non-squamous non-small cell lung cancer. Preclinical and clinical studies showed that pemetrexed had cytotoxic activity in many kinds of cancers including colorectal cancer. Erlotinib is a tyrosine-kinase inhibitor of EGFR, which was approved for the treatment of non-small cell lung cancer. Erlotinib also showed activity to colorectal cancer cells. Recently, Zhang et al. demonstrated synergistic cytotoxicity of pemetrexed and gefitinib in preclinical study.

In this multicenter, non randomized, open label phase II study, investigators aimed to evaluate the efficacy and safety of Pemetrexed and Erlotinib combination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 19 years
2. Histologic or cytologic confirmed diagnosis of colorectal carcinoma with metastatic (STAGE IV) disease.
3. Confirmed KRAS(codon 12 or 13) status
4. Prior chemotherapy for metastatic disease is required; prior regimens must include fluoropyrimidine, oxaliplatin and irinotecan
5. Eastern Cooperative Oncology Group performance status ≤ 2
6. Patients who can swallow oral medication.
7. Life expectancy of greater than 3 months
8. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1,500/mm3
   * hemoglobin ≥ 9 g/dl
   * platelets ≥ 100,000/mm3
   * serum total bilirubin ≤ 1.5 X institutional upper limit of normal
   * aspartate aminotransferase(SGOT)/alanine aminotransferase(SGPT) ≤ 3.0 X institutional upper limit of normal (≤ 5 times the upper institutional limits of normal if hepatic metastases are present)
   * serum creatinine ≤ 1.5 times the institutional upper limits of normal or Creatinine Clearance ≥ 50ml/min
9. The effects of Pemetrexed and Erlotinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because therapeutic agents used in this trial are known to be teratogenic, female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception (hormonal or barrier method of birth control; abstinence) during the study and for 6 months thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Participant is willing and able to give informed consent for participation in the study. Voluntary signed and dated written informed consent form in accordance with regulatory and institutional guidelines obtained before the performance of any protocol-related procedures not part of normal patient care.

Exclusion Criteria:

1. Previous treatment with Pemetrexed and Erlotinib
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pemetrexed or Erlotinib or other agents used in the study
3. Patients who can not allow the administration of Folic acid or Vitamin B12.
4. Past or current history of neoplasm other than colorectal carcinoma with a disease-free interval of less than 5 years, except for non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix.
5. Systemic chemotherapy within three weeks after the administration of the last before the test treatment
6. Major surgical operation or major trauma within 4 weeks.
7. Patients who have had wide-ranged radiotherapy within 4 weeks or limited radiotherapy within 2 2 weeks.
8. Persistent toxicity (> CTCAE grade 1) related to previous treatment except for the hair loss.
9. Patients with active brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Breast-feeding or pregnant female

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 2 years
Progression-free survival | up to 2 years

SECONDARY OUTCOMES:
Overall survival | up to 2 years
Disease control rate | up to 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joong Bae Ahn, Principal Investigator — Yonsei Cancer Center, Yonsei University Health System
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea